CLINICAL TRIAL: NCT02372552
Title: Clinical Evaluation of the Safety and Performance of Microwave Coagulation by the CROMA Electrosurgical System During Resection of Complex Colorectal Polyps
Brief Title: Microwave Coagulation Using CROMA Electrosurgical System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creo Medical Limited (Industry)
Collaborators: St Mark's Hospital, Harrow, UK (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML/014/001
Record Dates: First submitted 2015-02-10; First posted 2015-02-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-02

CONDITIONS: Polyp of Large Intestine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CROMA (Experimental): Microwave coagulation of small blood vessels
  Interventions: Device: CROMA

INTERVENTIONS:
Device: CROMA — Microwave coagulation of small blood vessels
  Other Names: Speedboat

SUMMARY:
This is a single centre, prospective, non-randomised pivotal clinical investigation to be undertaken at St Mark's Hospital, Harrow, UK.

DETAILED DESCRIPTION:
The study will recruit 30 patients undergoing endoscopic resection of complex colorectal polyps and be used to demonstrate safety and performance of the CROMA Electrosurgical System microwave coagulation modality. Study data will complement existing data to support a CE marking application for the CROMA Electrosurgical System (combined RF and microwave modalities).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age;
* After standard clinical work-up a benign appearing lower bowel lesion >2cm in diameter;
* Patient or authorised representative able to comprehend and sign the Informed Consent prior to enrolment in the study.

Exclusion Criteria:

* Aged <18 years of age;
* Pregnant or lactating females;
* Lower bowel lesions <2cm in diameter;
* Patients receiving regular systemic steroids;
* Patients who are immuno-compromised (either acquired or congenital);
* Patients with a known coagulopathy (either acquired or congenital);
* Patients on anti-platelet therapy at the time of the procedure, apart from low dose (75mg) aspirin alone;
* Concurrent participation in another experimental intervention or drug study;
* Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pre-coagulation of visible blood vessels and treatment of actively bleeding vessels, ≤1mm in diameter. | Peri-operative
  Performance will be assessed on the basis of number of vessels successfully coagulated.

SECONDARY OUTCOMES:
Safety: assessed using reported Adverse Events | 28 weeks
  Safety will be assessed using reported Adverse Events up to 28w post-operatively
Intra-operative complications | Intra-operative
  The proportion of patients with intra-operative complications will be reported
Post-procedural complications | 28 weeks
  The proportion of patients with post-procedural complications will be reported
Clinical outcome | 28 weeks
  The proportion of patients that go on to require further surgery during the immediate post-operative and follow up periods will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Brian Saunders, Professor, Principal Investigator — St. Mark's Hospital
Locations (1):
- Wolfson Unit for Endoscopy, St Mark's Hospital, Harrow, Middlesex, United Kingdom